CLINICAL TRIAL: NCT01374984
Title: Clinical Outcomes of VIGIV Treatment of Smallpox Vaccination Complications or Vaccinia Infection
Brief Title: VA-005 Clinical Outcomes of VIGIV Treatment of Smallpox Vaccination Complications or Vaccinia Infection
Status: Enrolling by invitation | Type: Observational
Sponsor: Emergent BioSolutions (Industry)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: VA-005
Record Dates: First submitted 2011-06-14; First posted 2011-06-17 (Estimated); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Complication of Smallpox Vaccination
Keywords: smallpox; vaccination; complications
MeSH Terms: conditions — Smallpox | interventions — human intravenous vaccinia immune globulin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A plasma sample for the determination of anti-vaccinia antibody level collected 5 days after VIGIV administration and 5 days after VIGIV re-dosing as well (if applicable). Samples collected Day 5 ±3 days will still provide valuable information for assessing anti-vaccinia antibody levels in these subjects post-VIGIV administration. While plasma samples are preferred, serum samples will also be accepted if available. Failure to obtain a Day 5 sample does not preclude retrospective enrollment into the VA-005 study to provide observational data only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects treated with VIGIV.: Subjects treated with VIGIV deployed from the US Strategic National Stockpile for any of the following conditions:
  * Eczema vaccinatum.
  * Progressive vaccinia.
  * Severe generalized vaccinia.
  * Vaccinia infections in individuals who have skin conditions.
  * Aberrant infections induced by vaccinia virus (except in cases of isolated keratitis).
  Interventions: Biological: VIGIV

INTERVENTIONS:
Biological: VIGIV — VIGIV is licensed in US, by the FDA, for the treatment of complications of smallpox vaccinations and is available to eligible patients regardless of participation in this study.
  Other Names: Vaccinia Immune Globulin Intravenous (Human)

SUMMARY:
This is a post-marketing study to verify the clinical benefits of VIGIV [CNJ-016, Vaccinia Immune Globulin Intravenous (Human), sterile solution] in the resolution of complications resulting from smallpox vaccination in eligible patients treated with VIGIV.

DETAILED DESCRIPTION:
This is an open-label Phase 4 study designed to collect additional data to assess the safety and efficacy of VIGIV [CNJ-016, Vaccinia Immune Globulin Intravenous (Human), sterile solution] in the first 100 consented patients treated with VIGIV.

ELIGIBILITY:
Inclusion Criteria:

Subjects treated with VIGIV deployed from the US Strategic National Stockpile for any of the following conditions:

* Eczema vaccinatum.
* Progressive vaccinia.
* Severe generalized vaccinia.
* Vaccinia infections in individuals who have skin conditions such as burns, impetigo, varicella-zoster, or poison ivy, or in individuals who have eczematous skin lesions because of either the activity or extensiveness of such lesions.
* Aberrant infections induced by vaccinia virus that include its accidental implantation in eyes (except in cases of isolated keratitis), mouth, or other areas where vaccinia infection would constitute a special hazard.
* Informed consent voluntarily signed by subject, legal guardian or representative to participate in the study. For minors, the informed consent form must be signed by a legally acceptable representative and when appropriate, informed consent/assent must also be obtained from the minor.

Exclusion Criteria:

None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who are administered VIGIV distributed from the US Strategic National Stockpile for the treatment of complications due to vaccinia vaccination or vaccinia infections.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Resolution of vaccinia infection complications | At hospital discharge (if not fully resolved at discharge then 1 month or 6 months as applicable)
  Change in number, size, type, and percentage of body affected by lesions following treatment.

SECONDARY OUTCOMES:
Vaccinia antibody levels | Day 5 post VIGIV-infusion
  Measurement of serum concentration of anti-vaccinia antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: David Cassie, MSc, Study Chair — Emergent BioSolutions

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: VIGIV [CNJ-016, Vaccinia Immune Globulin Intravenous (Human), sterile solution] United States Prescribing Information, 1/2010. — http://www.fda.gov/downloads/BiologicsBloodVaccines/BloodBloodProducts/ApprovedProducts/LicensedProductsBLAs/FractionatedPlasmaProducts/UCM199477.pdf